CLINICAL TRIAL: NCT01704313
Title: A Randonimised Trial Comparing Interrupted to Continuous Suturing Techniques in Radiocephalic Fistulae
Brief Title: A Trial of Interrupted vs Continuous Suturing Techniques for Radiocephalic Fistulae
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Emma Aitken (Other)
Responsible Party: Sponsor-Investigator, Emma Aitken, Clinical Research Fellow, Renal Surgery, NHS Greater Glasgow and Clyde
Organization: NHS Greater Glasgow and Clyde (Other)
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 12/WS/0089
Record Dates: First submitted 2012-10-08; First posted 2012-10-11 (Estimated); Last update posted 2012-10-11 (Estimated); Status verified 2012-10

CONDITIONS: End Stage Renal Failure
Keywords: Vascular access; Haemodialysis; Suturing technique
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Interrupted (Experimental): Interrupted suturing technique used around heel of anastomosis
  Interventions: Procedure: Interrupted
- Continuous (Active Comparator): Continuous suturing technique used for the anastomosis
  Interventions: Procedure: Continuous

INTERVENTIONS:
Procedure: Interrupted — Interrupted suturing technique used aroudn the heel of the vascular anastomosis
  Arms: Interrupted
Procedure: Continuous — Continuous suturing technique used for the anastomosis
  Arms: Continuous

SUMMARY:
Patients with end-stage renal failure require dialysis to remove toxins from their blood. Haemodialysis is best provided through a native arterio-venous fistula (AVF). Creation of an AVF requires a short (~1hr) surgical procedure to join the artery and vein together.

There are limited potential sites for fistula creation. Generally it is preferrable to utilise the most distal sites at the wrist first, as more proximal elbow procedures preclude subsequent use of the wrist should the initial fistula fail. The small diameter of artery and vein at the wrist requires precise surgical technique.

There are two potential techniques in common use for creating the arterio-venous anastomosis (the join between artery and vein) - continuous suturing and interrupted sutures. Whilst there are theoretical advantages to the interrupted technique, it is uncertain if these translate clinically into better success of creating the fistula. The aim of this study is therefore to compare the clinical success of the two techniques.

DETAILED DESCRIPTION:
The micro-vascular anastamosis required for creation of a radio-cephalic arteriovenous fistula, is technically challenging surgery. Primary patency rates for radiocephalic fistula varying between 50-75% in the literature and 60-95% within over own department. It is important to optimise primary patency rates as initial failure subjects the patient to risks of further surgery and often necessiates them commencing dialysis via a tunnelled line (which is less effective and associated with increased risks of infection) whilst a second attempt at creating a fistula is undertaken.

Multiple variations of both continuous and interrupted suture technique are described in the vascular literature, both in animal models of arterio-venous fistulae and in clinical studies in other specialities. However no study has compared the two techniques within clinical practice.

Evidence from in vivo animal studies is variable. Several authors have shown no difference in primary patency rates achieved with continuous suture versus interrupted suture technique used for anastomosis(Chen & Chen, 2001; Wilasrusmee et al 2007). Others have suggested that using a continuous suture causes a reduced cross-sectional area of the anastomosis compared to an interrupted technique (Tozzi & Hayoz, 2001). Similarly an interrupted suture technique permits expansion of the vessel at physiological pressures where as continuous technique does not (Norbert & Philip, 1996; Gerdisch & Hinkamp, 2003). This loss of compliance at the anastomosis can in turn lead to intimal hyperplasia, causing poor blood flow and failure of the anastamosis (Dorbin, 1994), indicating potential theoretical benefits of interrupted suturing.

There are no clinical studies comparing the two techniques and variation in practice varies considerably. The aim of this study therefore is the compare patency rates in radiocephalic fistulae by randomising to one or other anastomotic technique.

ELIGIBILITY:
Inclusion Criteria:

* End stage renal failure
* Undergoing surgery for creation of a radiocephalic fistula

Exclusion Criteria:

* Declines participation
* Unable to speak English or provide informed consent
* Radial artery diameter <1.8mm
* Cephalic wrist diameter at wrist <2mm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2012-05; Primary Completion 2013-08 (Estimated); Study Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
Primary patency | 6 weeks
  Primary patency is defined by the unequivocal presence of a thrill/ bruit and unassisted maturation a to permit dialysis

SECONDARY OUTCOMES:
Secondary patency | 6 weeks, 1 year
  Defined as assited patency to permit the fistula to be used for dialysis
Primary patency | 1 year
  Primary patency is defined as the unequivocal presence of thrill/ bruit and maturation of fistula so as to permit dialysis

CONTACTS AND LOCATIONS:
Overall Officials: David B Kingsmore, MBChB FRCS, Principal Investigator — NHS Greater Glasgow and Clyde
Locations (1):
- Department of Renal Surgery, Western Infirmary, Glasgow, United Kingdom

REFERENCES:
- [Derived] Aitken E, McColl G, Kingsmore D. The Role of Qutenza(R) (Topical Capsaicin 8%) in Treating Neuropathic Pain from Critical Ischemia in Patients with End-Stage Renal Disease: An Observational Cohort Study. Pain Med. 2017 Feb 1;18(2):330-340. doi: 10.1093/pm/pnw139. PMID 28204726